CLINICAL TRIAL: NCT05342207
Title: Endoscopic Plantar Fascia Release in Cases of Chronic Resistant Plantar Fasciopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mohamed Saeed Hamdy, Orthopedic surgery resident at sohag university, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-22-03-06
Record Dates: First submitted 2022-03-16; First posted 2022-04-22 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: in Cases of Chronic Resistant Plantar Fasciopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- cases (Experimental)
  Interventions: Procedure: Endoscopic plantar fascia release in cases of chronic resistant plantar fasciopathy

INTERVENTIONS:
Procedure: Endoscopic plantar fascia release in cases of chronic resistant plantar fasciopathy — A medial portal will be developed 1cm away from the plantar skin along a vertical line passing through the posterior border of the medial malleolus with the foot in neutral position. A 5 mm cannula will be then introduced through the lateral portal over the trocar. Irrigation fluid will be then connected. A 30-degree 4.0 mm endoscope will be inserted inside the cannula. A 4.5 motorized incisor blade will be then used to debride the subcutaneous tissue until full visualization of the shiny fibers of the plantar fascia will be possible. A needle was inserted vertically through the heel skin to act as a land mark for the middle of the plantar fascia. A scalpel blade will then introduced through the medial portal to divide the full thickness of the medial half of the plantar fascia into two leaflets under direct visualization . The posterior leaflet will be then totally debrided using a motorized incisor blade . The tunnel will then be irrigated and stitches will be done.

SUMMARY:
The plantar fascia is a thick tissue band that connects the heel bone (the medial tubercle of the under surface of the calcaneus) to the metatarsophalangeal joints, forming the medial arch of the foot, which supports the foot during walking. Irritation and scarring of the plantar fascia is one of the most common causes of heel pain .

Plantar fasciopathy accounts for 11% to 15% of all foot disorders in both athletes and sedentary patients .

Although commonly referred to using incorrect nomenclature as plantar fasciitis ,it is degenerative process (i.e. fasciopathy).The etiology of plantar fasciopathy is not clear. It can result from irritation due to overstrain of the fascia, which induces mucoid degeneration The pathologic ﬁndings include degenerative tissue changes without inﬂammatory mediators .

The diagnosis of plantar fasciopathy is determined by the medical history and physical examination ﬁndings. Typically, patients present with heel pain during weight bearing , especially in the early morning and with the ﬁrst steps after a period of inactivity .

Patients will usually have tenderness around the site of the plantar aponeurosis . The pain can be reproduced by stretching the diseased plantar aponeurosis by passive hyperextension of the metatarsophalangeal joints .

Endoscopic plantar fasciotomy is a relatively new procedure, involves an endoscopic approach to the heel, allowing a plantar aponeurosis release to be performed with delicate instruments, minimal dissection, and immediate weight bearing

ELIGIBILITY:
Inclusion Criteria:

* Adults more than 18 years old presented by a single site heel pain with local pressure at the origin of plantar fascia on the medial Calcaneal tuberosity for one year, with failure of at least two lines of conservative treatment including:

Non-steroidal anti-inflammatory drugs (NSAIDs), Corticosteroid injections, physical therapy, exercise program (Achilles tendon and plantar fascia stretching exercises) and orthotic devices (heel cup, molded shoe insert or night splint) for at least 3 months.

Exclusion Criteria:

* Patients younger than 18 years.
* Patients who had a local infection or a metabolic disorder especially diabetes, generalized polyarthritis, sero-negative arthropathy, , tarsal tunnel syndrome.
* Patients with congenital anomalies e.g pesplanus, pescavus, limb length discrepancy, in-toeing, neuro-muscular disorders.
* Patients with an ipsilateral or contralateral vascular or neurological abnormalities, or malignancies.
* Recent trauma or foot and ankle deformity or fractures.
* Active anticoagulation therapy or bleeding disorders
* Patients who received a corticosteroid injection within the previous four weeks.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-04 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
American Orthopedic Foot and Ankle-Hind foot Scale | 6 months following operation
  * Pain
  * Function
  * Alignment assessment

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Cottom JM, Maker JM, Richardson P, Baker JS. Endoscopic Debridement for Treatment of Chronic Plantar Fasciitis: An Innovative Technique and Prospective Study of 46 Consecutive Patients. J Foot Ankle Surg. 2016 Jul-Aug;55(4):748-52. doi: 10.1053/j.jfas.2016.02.005. Epub 2016 Apr 5. PMID 27066869
- [Background] Lui TH. Endoscopic Decompression of the First Branch of the Lateral Plantar Nerve and Release of the Plantar Aponeurosis for Chronic Heel Pain. Arthrosc Tech. 2016 Jun 6;5(3):e589-94. doi: 10.1016/j.eats.2016.02.018. eCollection 2016 Jun. PMID 27656382
- [Background] Oliva F, Piccirilli E, Berardi AC, Frizziero A, Tarantino U, Maffulli N. Hormones and tendinopathies: the current evidence. Br Med Bull. 2016 Mar;117(1):39-58. doi: 10.1093/bmb/ldv054. Epub 2016 Jan 19. PMID 26790696
- [Background] Sabir N, Demirlenk S, Yagci B, Karabulut N, Cubukcu S. Clinical utility of sonography in diagnosing plantar fasciitis. J Ultrasound Med. 2005 Aug;24(8):1041-8. doi: 10.7863/jum.2005.24.8.1041. PMID 16040817